CLINICAL TRIAL: NCT03144934
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose Study to Evaluate the Safety and Tolerability of GX-I7 in HPV-infected Female Volunteers
Brief Title: Safety and Tolerability of GX-I7 in HPV-infected Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GX-I7M-HPV-002
Record Dates: First submitted 2017-04-18; First posted 2017-05-09 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Human Papillomavirus
Keywords: HPV
MeSH Terms: interventions — efineptakin alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Administraion of investigational product (Experimental): * 0.25mg, 1mg, 3mg, 6mg, or 9mg (optional) of GX-I7
  * 6 subjects per each cohort
  * twice administration with 4-week intervals
  Interventions: Drug: GX-I7
- Administraion of placebo (Placebo Comparator): * GX-I7 vehicle (formulation buffer)
  * 2 subjects per each cohort
  * twice administration with 4-week intervals
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GX-I7 — Interleukin-7 (IL-7) is T cell growth factor that can be used for treating lymphopenia patients. GX-I7 is a protein drug recombining human IL-7 and hybrid Fc (hyFc). HyFc made by Genexine is composed of hinge-CH2 region of Immunoglobulin D (IgD) and CH2-CH3 region of Immunoglobulin G4 (IgG4). The recombined region is not exposed and each region's characteristics can reduce immunogenicity and improve the efficacy of drug. Consequently, it will be able to treat the patients with lymphopenia in effective ways.
  Other Names: IL-7-hyFc
  Arms: Administraion of investigational product
Drug: Placebo — This is the placebo of GX-I7 described above.
  Other Names: GX-I7 vehicle (formulation buffer)
  Arms: Administraion of placebo

SUMMARY:
This is a phase 1, randomized, double-blind, placebo-controlled, multiple ascending dose study to evaluate the safety and tolerability of GX-I7 in HPV-infected female volunteers

DETAILED DESCRIPTION:
The subjects who are adequately eligible to attend this clinical trial via screening will be assigned to four cohorts (five if necessary) and administered a single dose of GX-I7 solution or placebo drug for intravaginal injection at the visit 3 (Day0) and 7 (Day28). After completing scheduled tests at the visit 6 (Day 14), safety-related data of each cohort will be evaluated by Independent Safety Monitoring Committee (SMC). Dose escalation will proceed under the principal investigator, medical monitor, and the sponsor's mutual approval, referring to SMC's evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Subject willing and able to give informed consent
* Must be ≥19 and ≤45 years diagnosed with HPV infection in two tests within screening periods or have history of HPV infection within 6 months and diagnosed with HPV infection in one test within screening periods
* No clinical abnormality from ECG test
* Must agree to use appropriate contraceptive methods (ie, condoms, cervical cap in conjunction with spermicide, sterilization, and intra uterine device) during the study and for 3 months after the last dose of study drug.

Exclusion Criteria:

* Subject with HSIL or more severe HPV infection
* History of a known or suspected hypersensitivity, shock, or past history to the investigational drug or to similar drugs
* Malignant tumor within 5 years other than successfully treated skin cancer that is not melanoma
* Active infection or history of infection that required intravenous injection of antibiotics 4 weeks prior to the first administration of the investigational drug
* Female subject unwilling to stop breastfeeding or pregnancy
* Positive result from serology examination for human immunodeficiency virus (HIV)
* Major surgery within 3 months other than access surgery
* Mental disorder or other central nervous system disorder determined that the study evaluation cannot be conducted
* Participation in any clinical study within 30 days
* History of alcohol or drug abuse within 6 months prior to the screening
* Any other ineligible condition at the discretion of the investigator that would be ineligible to participate the study

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the safety of GX-I7 compared to placebo. | 12 weeks
  Local and systemic adverse events will be assessed by Department of AIDS (Table for Grading the Severity of Adult and Pediatric Adverse Events, 2004) and Toxicity Grading Scale for Healthy Volunteers Enrolled in Preventive Vaccine Clinical Trials, respectively. Also, vital signs (blood pressure, heart rate, and body temperature), physical examination, laboratory tests, upper abdomen ultrasound, immunogenicity test, and concentration of the investigational drug in blood sample will be assessed throughout the screening and study period.

SECONDARY OUTCOMES:
Type of Humanpapillo Virus (HPV) Persistent Infection of Human Papilloma Virus (HPV) | at week 0 (Day 0) and week 4 (Day 28)
  Perform liquid-based cytology after each injections

CONTACTS AND LOCATIONS:
Overall Officials: Jae Kwan Lee, MD, PhD, Principal Investigator — Korea University Guro Hospital
Locations (4):
- South Korea (4):
  - Chungnam National University Hospital, Daejeon
  - Yonsei University Health System, Severance Hospital, Seoul
  - Hallym University Medical Center-Kangnam, Seoul
  - Korea University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No